CLINICAL TRIAL: NCT03664947
Title: The Impact of Video Based Game Exercise Approaches on Sleep in Children With Acute Lymphoblastic Leukemia: Randomized Single Blind Controlled Study
Brief Title: The Impact of Exercise Approaches on Sleep in Children With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BezmialemVUFBC
Record Dates: First submitted 2018-07-13; First posted 2018-09-11 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Oncology Problem; Sleep
Keywords: exercise; sleep problems; acute lymphoblastic leukemia
MeSH Terms: conditions — Motor Activity; Parasomnias; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Experimental): The exergaming training programs have included recent daily living activities in games. In our study we have planned the Nintendo Wii Fit Plus Game Console in the therapy training.
  Interventions: Other: exercise
- control (No Intervention): No exercise training applied for the control group.

INTERVENTIONS:
Other: exercise — After the initial evaluations, a video-based gaming console exercise program will be implemented for 8 weeks, taking into account the possibility of accepting and participating in treatment with children. Exercises applied by a Nintendo Wii Fit Plus System. Evaluations will be repeated at the end of treatment.
  Arms: exercise

SUMMARY:
Sleep is one of the basic and indispensable daily life activities that affect the quality of life and health of individuals and is a concept with physiological, psychological and social dimensions. In the literature, sleep difficulties and problems have begun to be investigated in children with acute lymphoblastic leukemia and have not been found in national publications. In these children, sleep quality, strengths and disorders and a study evaluating this variation on a scale have not been found. For this reason, our study will be done in order to determine the factors affecting sleep and sleep in children with cancer and to show the effect of exercise on these factors.

DETAILED DESCRIPTION:
Primeraly that progresses in the disease process, secondary problems seen with the effects of symptoms make it difficult to cope with disease and treatment process in children with acute lymphoblastic leukemia (ALL) . Sleep difficulty is not affected by the direct effects of the disease but it is affected and becomes more difficult with the fatigue and difficulty of treatment as a secondary. Parents with ALL children stated that they experienced 12.4% of sleeping difficulty. It turns out that about a quarter of the children are sleeping problems. It is stated that 27% of these children have drowsiness, and more than 25% of them have frequent awakenings at night. It is also stated that parents use the option of rest-sleep as an option to benefit from treatment in coping with the disease, but children with sleeping difficulties also make it difficult to treat them. Being a healthcare professional as a biopsychosocial approach model and planning the treatment interventions for the deficiencies and disorders that will be done in order to get rid of the symptoms of the disease as soon as possible will make it easier to cope with the disease with both child and parent and multidisciplinary approach. In this way, we will investigate the effects of children's exercise habits on their sleep and sleep related complaints by using video-based game consoles which are currently used in our workout approaches. The games to be selected from the aerobic exercise programs that are used to increase the functional capacity on the basis of exercise will also be targeted to the exercises with maximum motivation and participation of the children. In the exercises where goodness and continuity are also taken into consideration, in-game guidance will be provided with verbal commands under the supervision of a physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Having ALL a diagnosis
* Being between 2-18 years of age
* Therapy (surgery, chemotherapy, radiotherapy) to be finished

Exclusion Criteria:

* Continue active treatment (surgery, chemotherapy, radiotherapy)
* Recurrence of the disease
* Any mental / physical problem that will have a cooperative problem

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Polysomnography, Characteristics of Sleep | 12 weeks
  Polysomnography is used increasingly to investigate patients with possible sleep apnoea/ hypopnoea syndrome. It is a report that which indicate sleep quality.

SECONDARY OUTCOMES:
Childhood Sleep Habit Questionnaire (CSHQ) | 12 weeks
  The CSHQ is a parent-rated questionnaire comprised of 45 items; 33 scored questions, and 7 additional items intended to provide other relevant information pertaining to sleep behavior. Each scored question is rated on a 3-point scale as occurring "usually", "sometimes", or "rarely". A number of items on the questionnaire are reverse-scored, so that higher scores consistently indicate problem behaviors. Ratings are combined to form eight subscales: Bedtime Resistance, Sleep Onset Delay, Sleep Duration, Sleep Anxiety, Night Wakings, Parasomnias, Sleep Disordered Breathing, and Daytime Sleepiness. A Total Sleep Disturbances score is calculated as the sum of all CSHQ scored questions, and can range from 33 to 99. A Total Sleep Disturbances score of over 41 indicates a pediatric sleep disorder, as this cutoff has been shown to accurately identify 80% of children with a clinically diagnosed sleep disorder.
Epworth Sleepiness Scale (ESS) | 12 weeks
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'. The questionnaire takes no more than 2 or 3 minutes to answer.
Pitsburg Sleep Quality Index (PSQI) | 12 weeks
  The Pitsburg Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No